CLINICAL TRIAL: NCT03115918
Title: Randomized Trial Examining the Impact of Pancreatic Duct Stent Placement in Patients With Acute Necrotizing Pancreatitis in the Prevention of Walled-off Necrosis
Brief Title: Pancreatic Duct Stent for Acute Necrotizing Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 922733
Record Dates: First submitted 2017-01-17; First posted 2017-04-14 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Necrotizing Pancreatitis; Walled Off Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pancreatic Duct Stent Placement (Active Comparator): Subject will have placement of either the Advanix or Cook Pancreatic Stent placed.
  Interventions: Device: Pancreatic Duct Stent Placement
- No Pancreatic Duct Stent Placement (Active Comparator): Subject will not have a pancreatic Duct stent placed.
  Interventions: Other: No Pancreatic Duct Stent Placement

INTERVENTIONS:
Device: Pancreatic Duct Stent Placement — Patients will be randomly allocated to either treatment arm to have a PD stent placed.
  Arms: Pancreatic Duct Stent Placement
Other: No Pancreatic Duct Stent Placement — Patients will be randomly allocated to either treatment arm and not receive PD placement.
  Arms: No Pancreatic Duct Stent Placement

SUMMARY:
The research design is a randomized prospective clinical study comparing the incidence of Walled Off Necrosis (WON) in patients with acute necrotizing pancreatitis.

DETAILED DESCRIPTION:
This is a randomized trial comparing the incidence of WON in patients with acute necrotizing pancreatitis, according to the placement or non-placement of an Advanix or a Cook Pancreatic Duct (PD) stent during Endoscopic Retrograde Cholangiopancreatography (ERCP) within 1-2 week of symptom onset. Patients will be randomly allocated to either treatment arm i.e. to either PD stent placement or no PD placement in a 1:1 ratio. The type of stent to be placed is at the discretion of the physician based on the clinical needs and presentation of the patient at the time of procedure. This is based on factors such as the size of the WON, the patient's anatomy, and other variables. Patients will be assessed at 4-6 weeks post-ERCP for the primary outcome measure, which is the incidence of WON on contrast-enhanced CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years
2. The subject (or when applicable the subject's LAR) is capable of understanding and complying with protocol requirements.
3. The subject (or when applicable the subject's LAR) is able to understand and willing to sign an informed consent form prior to the initiation of any study procedures.
4. All patients with acute necrotizing pancreatitis and bedside index for severity in acute pancreatitis (BISAP) score of ≥ 3, who have been referred to Florida Hospital for Percutaneous endoscopy gastrojeunostomy (PEG-J) tube placement and/or ERCP for assessment of the PD
5. Absence of pancreatic fluid collection (defined as those > 3cm in size located along the course of the main PD on cross-sectional imaging) at the time of study enrollment
6. No disconnected pancreatic duct syndrome (DPDS) on cross-sectional imaging or ERCP

Exclusion Criteria:

1. Age <19 years
2. Unable to obtain consent for the procedure from either the patient or LAR
3. Patients with acute interstitial pancreatitis, without pancreatic necrosis
4. Patients with BISAP score ≤ 2
5. Patients with pancreatic fluid collection > 3cm in size located along the course of the main PD on cross-sectional imaging prior to the initial ERCP
6. Patients with DPDS on cross-sectional imaging or ERCP
7. Unable to safely undergo ERCP for any reason
8. Failed cannulation during ERCP

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Incidence of WON between the PD stent and no PD stent groups | 4-6 weeks post-index ERCP
  The primary aim of the study is to compare the incidence of WON between the PD stent and no PD stent groups at 4-6 weeks post-index ERCP.

SECONDARY OUTCOMES:
Rates of WON Intervention | 6 weeks
  Incidence of WON requiring intervention of any type (including endoscopic, surgical or interventional radiology interventions)
Rates of DPDS | 6 weeks
  Incidence of DPDS, as determined by ERCP or Magnetic Resonance Cholangiopancreatography (MRCP)
Number of patients with Adverse events | 6 weeks
  Incidence of procedure related adverse events
Rates of additional interventions resulting from complications | 6 weeks
  Incidence of other interventions undertaken as clinically indicated for complications of acute pancreatitis
Number of patients with Acute pancreatitis | 6 weeks
  Clinical adverse events related to underlying acute pancreatitis
Number of patients with Local complications | 6 weeks
  Clinical adverse events arising as a result of local complications of acute pancreatitis
Number of patients with Systemic complications | 6 weeks
  Clinical adverse events arising as a result of systemic complications of acute pancreatitis
Length of stay | 6 weeks
  Duration of hospitalization in days
Cost | 6 weeks
  Total hospital costs in US Dollars

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.

REFERENCES:
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Freeman ML, Werner J, van Santvoort HC, Baron TH, Besselink MG, Windsor JA, Horvath KD, vanSonnenberg E, Bollen TL, Vege SS; International Multidisciplinary Panel of Speakers and Moderators. Interventions for necrotizing pancreatitis: summary of a multidisciplinary consensus conference. Pancreas. 2012 Nov;41(8):1176-94. doi: 10.1097/MPA.0b013e318269c660. PMID 23086243
- [Background] Garg PK, Madan K, Pande GK, Khanna S, Sathyanarayan G, Bohidar NP, Tandon RK. Association of extent and infection of pancreatic necrosis with organ failure and death in acute necrotizing pancreatitis. Clin Gastroenterol Hepatol. 2005 Feb;3(2):159-66. doi: 10.1016/s1542-3565(04)00665-2. PMID 15704050
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Nadkarni NA, Kotwal V, Sarr MG, Swaroop Vege S. Disconnected Pancreatic Duct Syndrome: Endoscopic Stent or Surgeon's Knife? Pancreas. 2015 Jan;44(1):16-22. doi: 10.1097/MPA.0000000000000216. PMID 25493375
- [Background] van Santvoort HC, Besselink MG, Bakker OJ, Hofker HS, Boermeester MA, Dejong CH, van Goor H, Schaapherder AF, van Eijck CH, Bollen TL, van Ramshorst B, Nieuwenhuijs VB, Timmer R, Lameris JS, Kruyt PM, Manusama ER, van der Harst E, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, van Leeuwen MS, Buskens E, Gooszen HG; Dutch Pancreatitis Study Group. A step-up approach or open necrosectomy for necrotizing pancreatitis. N Engl J Med. 2010 Apr 22;362(16):1491-502. doi: 10.1056/NEJMoa0908821. PMID 20410514
- [Background] Casas M, Mora J, Fort E, Aracil C, Busquets D, Galter S, Jauregui CE, Ayala E, Cardona D, Gich I, Farre A. [Total enteral nutrition vs. total parenteral nutrition in patients with severe acute pancreatitis]. Rev Esp Enferm Dig. 2007 May;99(5):264-9. doi: 10.4321/s1130-01082007000500004. Spanish. PMID 17650935
- [Background] Gupta R, Patel K, Calder PC, Yaqoob P, Primrose JN, Johnson CD. A randomised clinical trial to assess the effect of total enteral and total parenteral nutritional support on metabolic, inflammatory and oxidative markers in patients with predicted severe acute pancreatitis (APACHE II > or =6). Pancreatology. 2003;3(5):406-13. doi: 10.1159/000073657. Epub 2003 Sep 24. PMID 14526151
- [Background] Louie BE, Noseworthy T, Hailey D, Gramlich LM, Jacobs P, Warnock GL. 2004 MacLean-Mueller prize enteral or parenteral nutrition for severe pancreatitis: a randomized controlled trial and health technology assessment. Can J Surg. 2005 Aug;48(4):298-306. PMID 16149365
- [Background] Petrov MS, Kukosh MV, Emelyanov NV. A randomized controlled trial of enteral versus parenteral feeding in patients with predicted severe acute pancreatitis shows a significant reduction in mortality and in infected pancreatic complications with total enteral nutrition. Dig Surg. 2006;23(5-6):336-44; discussion 344-5. doi: 10.1159/000097949. Epub 2006 Dec 12. PMID 17164546
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Yi F, Ge L, Zhao J, Lei Y, Zhou F, Chen Z, Zhu Y, Xia B. Meta-analysis: total parenteral nutrition versus total enteral nutrition in predicted severe acute pancreatitis. Intern Med. 2012;51(6):523-30. doi: 10.2169/internalmedicine.51.6685. Epub 2012 Mar 15. PMID 22449657
- [Background] Varadarajulu S, Noone T, Hawes RH, Cotton PB. Pancreatic duct stent insertion for functional smoldering pancreatitis. Gastrointest Endosc. 2003 Sep;58(3):438-41. doi: 10.1067/s0016-5107(03)00025-7. PMID 14528225
- [Background] Lau ST, Simchuk EJ, Kozarek RA, Traverso LW. A pancreatic ductal leak should be sought to direct treatment in patients with acute pancreatitis. Am J Surg. 2001 May;181(5):411-5. doi: 10.1016/s0002-9610(01)00606-7. PMID 11448431
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Varadarajulu S, Rana SS, Bhasin DK. Endoscopic therapy for pancreatic duct leaks and disruptions. Gastrointest Endosc Clin N Am. 2013 Oct;23(4):863-92. doi: 10.1016/j.giec.2013.06.008. Epub 2013 Jul 12. PMID 24079795